CLINICAL TRIAL: NCT05419284
Title: Feasibility of the Geriatric Activation Program Pellenberg With the Informal Caregiver as Exercise Partner of the Physiotherapist (GAPP+Care)
Brief Title: Feasibility of the Geriatric Activation Program Pellenberg With Caregiver Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Margaretha van Dijk, Principal Investigator, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S66154
Record Dates: First submitted 2022-05-18; First posted 2022-06-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Hip Fractures; Stroke; Frailty
Keywords: geriatric patients; geriatric rehabilitation; physiotherapy; caregiver involvement
MeSH Terms: conditions — Hip Fractures; Stroke; Frailty

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient (Experimental): GAPP+Care
  Interventions: Other: GAPP+Care
- caregiver (Experimental): +Care
  Interventions: Other: +Care
- healthcare professional of the ward (Other): observation of GAPP+Care
  Interventions: Other: Observation of GAPP+Care

INTERVENTIONS:
Other: GAPP+Care — standard physiotherapy 45 minutes per day, 5 day a week (GAPP)
  + 3 extra exercise sessions led by a caregiver (+Care)
  Arms: patient
Other: +Care — 3 extra exercise moments led by a caregiver: one physiotherapist-caregiver-patient exercise session: the physiotherapist will educate and train the caregiver on the exercises and hands-on skills.
  Two caregiver-patient exercise sessions
  Arms: caregiver
Other: Observation of GAPP+Care — Healthcare workers in the geriatric rehabilitation ward will be interviewed on their opinions on GAPP+Care
  Arms: healthcare professional of the ward

SUMMARY:
This interventional study aims to see if involving caregivers as exercise partners with the physiotherapist throughout in-hospital geriatric rehabilitation and the first six weeks following discharge is feasible.

Caregivers will receive hands-on training from physiotherapists so that they can assist their family members with their exercises. The caregivers will provide 30-minute exercise sessions three times each week in addition to the standard physiotherapy.

The researchers want to know how many people are eligible for GAPP+CARE and how willing they are to participate. The researchers also want to know about the program's hindering and facilitating elements, as well as its fidelity and retention rate. Apart from that, the researchers want to examine if an effectiveness study and the used outcome measures are viable.

DETAILED DESCRIPTION:
To meet the WHO guideline for daily exercise during and after hospitalization, physiotherapists must find ways for geriatric patients to be active outside of therapy time. Geriatric patients require assistance or supervision to exercise safely, yet physiotherapists and nurses are short on time. Instead, by providing carers with tools and instruction, the researchers might turn them into exercise partners for the physiotherapist.

The investigators designed an exercise program (GAPP+Care) customized to the caregiver's ability to exercise safely with their loved one, based on the ideas and exercises of our standard physiotherapy program, the Geriatric Activation Program Pellenberg (GAPP). Through semi-structured interviews, patients and their caregivers were involved in developing and validating GAPP+Care, including the exercise booklet.

GAPP+Care consists of GAPP (the usual physiotherapy treatment) and three additional 30-minute exercise sessions with the caregiver each week (+Care). +Care will continue at home for the first six weeks after discharge, and GAPP will be replaced with physiotherapy performed by a private physiotherapist, as described at discharge (a prescription for home physiotherapy 3 times a week, for 60 sessions F-pathology or 18 sessions).

The initial +Care session is with a ward physiotherapist who will show the caregiver how to utilize the GAPP+Care handbook and the exercises and teach them how to support the patient during the exercises. During hospitalization, one of the three weekly sessions will be led by a ward physiotherapist to reinforce the hands-on skills and knowledge. These physiotherapy-patient-caregiver sessions will consist of two home visits and four phone calls after the patient has been discharged.

The goal of this exploratory study is to see if GAPP+Care is feasible. The researchers want to know how many people are eligible and how willing they are to participate. The researchers also want to assess the program's hindering and facilitating elements, as well as its fidelity and retention rate. Aside from that, the researchers want to evaluate if an effectiveness study and the used outcome measures are viable.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Patients from geriatric rehabilitation unit, with various pathologies
* ≥ 70 years old
* ≥ 10m of walking with walking aid and under supervision
* Berg Balance Scale (BBS) < 30/56
* Medically stable as determined by the attending physician
* Expecting at least 3 weeks of rehabilitation

Exclusion Criteria:

* No available caregiver
* Unable to understand instructions

Caregivers:

Inclusion Criteria:

* A person who is willing to support the patient in performing exercises at least 3 times a week for 30 minutes. An informal carer is defined as an unpaid member of a person's social network who helps the patient with activities of daily living.

Exclusion Criteria:

* Physical unable to support the patient
* Unable to understand instructions

Healthcare providers

Inclusion Criteria:

* Someone who works on our ward, comes into contact with patients and may experience GAPP+CARE or its effects; nurse, physiotherapist, occupational therapist, social worker, doctor, logistical worker.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible individuals and their willingness to participate in GAPP+Care | 1 year
  Number of available patients on the ward and number of eligible patients and caregivers and number of patients and caregivers who participate

SECONDARY OUTCOMES:
Feasibility, appropriateness, and the hindering and facilitating factors of GAPP+Care | patients and caregivers 2 times (at day of discharge and at the end of week 6 after discharge), healthcare providers 1 time (in the last 6 months of the study)
  Semi-structured interviews with patients, caregivers and healthcare providers
Fidelity to GAPP+Care | up to 12 weeks
  Number of exercise moments with physiotherapist; Noted in exercise diary Number of exercise moments with caregiver; Exercise Diary Number and kind of exercises with caregiver; Exercise Diary
Retention rate of participants | 1 year
  Number of dropouts
Number of falls during the +Care sessions | up to 12 weeks
  number of falls noted in the exercise diary or mentioned during the interviews
Private physiotherapy after discharge | 6 weeks
  number of sessions per week
Use of the activity monitor MOX, Maastricht Instruments | first week at baseline, first week after discharge (starting at day of discharge), and week 6 after discharge
  measuring daily activity in minutes/24hours (sedentary - standing - dynamic)
Functional balance | 3 times over 10 weeks: baseline, at day of discharge (up tot 6 weeks after baseline) and at end of week 6 after discharge
  Berg Balance Scale (BBS) 0-56, a higher score means a better outcome
Hand squeeze force | 3 times over 10 weeks: baseline, at day of discharge (up tot 6 weeks after baseline) and at the end of week 6 after discharge
  Maximum handgrip with dominant hand, measured with the Martin Vigory dynamometer, in kPa
Walking speed | 3 times over 10 weeks: baseline, at day of discharge (up tot 6 weeks after baseline) and at the end of week 6 after discharge
  4m walking test (4mWT), m/s
Quality of life patient and caregiver | 3 times over 10 weeks: baseline, at day of discharge (up tot 6 weeks after baseline) and at end of week 6 after discharge
  Visual analog scale of quality of life (VAS QoL), 0-10 a higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johan Flamaing, PhD, MD, Principal Investigator — KU UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided